CLINICAL TRIAL: NCT06586710
Title: Interferon Pathway Activation in Monogenic and Non-monogenic Forms of Pediatric SLE With Renal Involvement. Multicenter Observational Study of Biological Samples.
Brief Title: Interferon Pathway Activation in Monogenic and Nonmonogenic Forms of Pediatric SLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Carmela Errichiello, Principal Investigator, Meyer Children's Hospital IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NEFRO-LES
Record Dates: First submitted 2024-02-20; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Systemic Lupus Erythematosus of Childhood

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Activation of interferon pathway (Other): Assessment activation of interferon pathway on biological samples (blood and kidney biopsy) in cSLE patients
  Interventions: Other: Assessment activation of interferon pathway

INTERVENTIONS:
Other: Assessment activation of interferon pathway — * Peripheral blood collection (as part of routine blood draws) on which interferon signature will be performed at the time of enrollment and in case of remission and/or any renal flare.
  * Renal biopsies (routinely performed for diagnostic purposes and during clinical follow-up) on which Myxovirus resistance protein 1 (MXA) expression and histopathologic characterization will be assessed.
  * Collection of clinical and laboratory data from routine visits performed at baseline and 3, 6, 12, and 24 months (or last available visit) after the renal biopsy was performed.

SUMMARY:
Pediatric SLE includes monogenic forms, some of which involve the interferon type I (IFN-I) pathway. The IFN-I pathway is renally active in adult SLE and correlates with the extent of renal damage. In pediatric SLE, and particularly in lupus nephritis, activation of the IFN-I pathway has never been studied, nor is it known whether monogenic forms underlie more pronounced interferon activation.

DETAILED DESCRIPTION:
Pediatric systemic lupus erythematosus (SLE) (cSLE), compared with adult SLE, is characterized by a more severe phenotype, with more marked hematologic, neuropsychiatric, and renal changes. Lupus nephritis is a pivotal manifestation of pediatric SLE and an important prognostic factor. It is hypothesized that activation of the interferon pathway is more pronounced in monogenic forms, in which the response to IFN-I represents the primary alteration and likely the main pathogenic mechanism.

This finding may also be relevant in light of the availability of new drugs that selectively target the IFN-I pathway.

Demonstration of IFN-I pathway activation could be used as a diagnostic algorithm in aggressive pediatric forms resistant to immunosuppressive therapy and represent a therapeutic target.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SLE arising before the age of majority (until the age of 18 years) according to SLICC and/or EULAR criteria 2019;
* Clinical, laboratory and/or histologic evidence of renal involvement manifested before the age of 18 years;
* Signature of informed consent.

Exclusion Criteria:

* Onset of renal disease after the age of 18 years;
* SLE secondary to drugs or associated with other diseases such as systemic sclerosis, rheumatoid arthritis, Sjögren's syndrome, and other connectivities.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference between monogenic and non-monogenic forms of cSLE | At the enrollment, in case of renal flare, in case of disease remission
  Quantification of the IFN-I target genes distinguishing between monogenic and non-monogenic forms.
Evaluation of expression of MXA protein in renal biopsy | Biopsy available at enrollment
  Evaluation of expression of MXA protein in renal biopsy (by fluorescence microscopy), distinguishing between genetic and non-genetic forms
Evaluation of the proportions of the various WHO histological classes of renal biopsy | At the end of the study (24 months after enrollment)
  Evaluation of the proportions of the various WHO histological classes of renal biopsy in patients with monogenic and non-monogenic lupus nephritis.
  Histological diagnosis at renal biopsy: WHO histological pattern, activity index, chronicity index, renal TMA

SECONDARY OUTCOMES:
Phenotype characterization of cSLE | At the onset of the disease, 3, 6, 12, 24 months from the kidney biopsy,
  Description of clinical parameters, as SLEDAI-2K, in patients with cSLE and renal involvement, distinguishing between monogenic and non-monogenic forms.
  Description of laboratory parameters as renal function (eGFR CKiD 25) in patients with cSLE and renal involvement, distinguishing between monogenic and non-monogenic forms
Correlation between the clinical phenotype, response to treatment and amplification of the interferon pathway | At the onset of the disease, 3, 6, 12, 24 months from the kidney biopsy,
  Correlation between the clinical phenotype (laboratory parameters and during renal flare), response to treatment and amplification of the interferon pathway, distinguishing between monogenic and non-monogenic forms.
  Clinical, laboratory and histological data relating to any renal flare: number of flares, date of the flare, months from the first biopsy diagnosis of lupus nephritis, clinical manifestations, data from the biopsy performed during the flare, WHO histological pattern compared with the first biopsy, activity index, chronicity index, induction therapy, maintenance therapy

CONTACTS AND LOCATIONS:
Overall Officials: Carmela Errichiello, Principal Investigator — Meyer Children's Hospital IRCCS, Florence, Italy
Locations (3):
- Italy (3):
  - Meyer Children's Hospital IRCCS, Florence
  - IRCCS Gianna Gaslini, Genova
  - IRCCS Humanitas Research Hospital, Rozzano

IPD SHARING:
Plan to Share IPD: No